CLINICAL TRIAL: NCT02203097
Title: The Effect of Different End-tidal Carbon-dioxide Levels on Cerebral CO2 Vasoreactivity and the Stiffness of Systemic Arteries During Propofol Anesthesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Debrecen (Other)
Responsible Party: Principal Investigator, Tamas Vegh, MD, assistant lecturer anesthesiologist and intensive care specialist, University of Debrecen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 030167-006/2014/OTIG; 2345 (Other: University of Debrecen, RKEB/IKEB)
Record Dates: First submitted 2014-07-25; First posted 2014-07-29 (Estimated); Last update posted 2017-03-09 (Actual); Status verified 2017-03

CONDITIONS: Propofol-anaesthesia Via Target-controlled Infusion
Keywords: Target controlled infusion; propofol; cerebral vasoreactivity; arterial stiffness; Transcranial Doppler; SphygmoCor
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Propofol (Experimental): Propofol is administered to all patients via target-controlled infusion (TCI) to reach 4 mcg/ml constant plasma concentration according to the Schneider model during the course of the narcosis.
  Interventions: Procedure: Partial pressure of CO2 at the end of an exhaled breath; Drug: Propofol

INTERVENTIONS:
Procedure: Partial pressure of CO2 at the end of an exhaled breath — Three previously defined EtCO2 levels (partial pressure of CO2 at the end of an exhaled breath) were adjusted during anesthesia.
  Other Names: EtCO2
Drug: Propofol — Propofol is administered to all patients via target-controlled infusion (TCI) to reach 4 mcg/ml constant plasma concentration according to the Schneider model during the course of the narcosis.
  Other Names: Diprivan

SUMMARY:
Purpose:

The purpose of this study is to examine the effect of different carbon-dioxide concentrations on cerebral CO2 sensitivity and the resistance and stiffness of systemic arteries during anesthesia with target-controlled infusion anesthesia using intravenous propofol. Propofol is a widely and commonly used intravenous anaesthetic, that is mainly used for the induction of general anesthesia and the maintenance of total intravenous anaesthesia (TIVA).

Changes in the velocity of cerebral blood flow and arterial stiffness due to the different exhaled carbon-dioxide concentrations will allow us to conclude how propofol affects these parameters during the course of the narcosis.

Instruments:

An ultrasound device called transcranial doppler (TCD) is used to measure the velocity of blood flow within a main artery located inside the skull.

A tonometry device named SphygmoCor is used to assess the pressure wave proceeding in the radial artery, from which the stiffness of the systemic vessels can be concluded.

Measurements:

- Examinations with the ultrasound and tonometry devices are carried out once before the operation, three times during the intervention, with different exhaled CO2 values and once after the operation is completed.

Hypothesis:

- Propofol alters cerebral carbon-dioxide sensitivity and the stiffness of systemic arteries during TCI anaesthesia.

DETAILED DESCRIPTION:
Study protocol:

- The study is conducted in four stages: in the first stage, measurements are performed preoperatively in awake patients. Patients are placed in supine position and mean arterial blood pressure (MAP), heart rate, oxygen saturation are measured. The transcranial doppler (TCD) probe is fixed in place by applying a headband to maintain a constant angle of insonation. Mean blood flow velocity (MBFV) and pulsatility index (PI) in the middle cerebral artery (MCA) are obtained. MCA is insonated through the right temporal window by using pulsed 2 megahertz TCD ultrasound probe. Identification of the MCA is confirmed by using standard criteria, at a depth of 45-55 mm. Cerebral CO2 vasoreactivity is calculated as the percentage change in MBFV or PI for mmHg change in end-tidal CO2 (ETCO2).

SphygmoCor is placed on the left radial artery to obtain data about the central aortic blood pressure, augmentation pressure (AP) and augmentation index normalised to a 75 beat per minute heart rate (Alx75). From the derived aortic pulse, calculations can be made, using the area under the systolic and diastolic part of the curve, to determine the heart's ratio of oxygen supply and demand, it is called the subendocardial viability ratio (SEVR).

As part of the premedication each patient receives 100 mg diclofenac per os 30 minutes and 500 ml Lactated-Ringer infusion 60 minutes prior to the operation.

Anesthesia is induced and maintained with target-controlled infusion anesthesia (TCI) using intravenous propofol at 4 mcg/ml constant plasma concentration. Analgesia is provided by using 2 ug/kg sufentanyl bolus dose at the time of induction. Afterwards 0.6 mg/kg rocuronium is given for muscle paralysis and subsequently patients were intubated with a suitable intratracheal tube. After induction of anaesthesia, the patients are placed on a mechanical ventilation system, using a volume-controlled setting with an air and oxygen mixture set to 0.4 fraction of inspired oxygen (FiO2) , the fresh gas flow rate to 2 l/min. .

Differences in the depth of anesthesia could influence cerebral activity, thereby cerebral metabolism and blood flow. Bispectral index is placed onto every patient in order to assure constant depth of anaesthesia during the intervention.

The second series of TCD and SphygmoCor measurements are performed 20 minutes after the respiratory rate is set to maintain end-tidal CO2 at 40 mmHg in order to allow sufficient time for equilibrium to be reached and the effect of drugs used for the induction of anesthesia to be terminated. Subsequently the examinations are repeated twice again at 35 and 30 mmHg ETCO2. The measurements were carried out 5-5 minutes after adjusting the minute ventilation to reach target ETCO2 values.

Statistical methods:

- Comparisons between the preoperative and three intraoperative stages of the study are made using repeated measures ANOVA with the Bonferroni post hoc correction. The relationship between MBFV, PI and ETCO2 is assessed using linear regression, while the connection between SEVR, pulse and Alx75 is calculated with bivariate correlation.

ELIGIBILITY:
Inclusion Criteria:

* Above the age 18
* American Society of Anesthesiologists (ASA) physical classification I. or II.
* Patients undergoing elective varicotomy, inguinal hernioplasty or breast surgery in general anesthesia

Exclusion Criteria:

* Patients with cerebral, cardiac or systemic vascular disorders (hypertension, diabetes)
* Patients receiving medication that affects the blood vessels (antihypertensive, antidiabetic, antiarrhythmic medications)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Blood flow velocity in the middle cerebral artery | Changes from baseline in blood flow velocity at the 15th, 20th and 25th minutes of the operation
  Systolic, diastolic and mean blood flow velocities are measured with transcranial doppler device.

SECONDARY OUTCOMES:
Arterial wall stiffness of the radial artery | Changes from baseline in arterial stiffness at the 15th, 20th and 25th minutes of the operation
  The stiffness of the radial artery is assessed. Stiffness rate is concluded from the augmentation pressure and augmentation index, from which both values are provided by the tonometry device.
Changes in the central systolic and diastolic blood pressure | Changes from baseline in central blood pressure at the 15th, 20th and 25th minutes of the operation
  Central blood pressure values are measured by means of tonometry device on the radial artery.

OTHER OUTCOMES:
Changes in subendocardial viability ratio (SEVR) | Changes form baseline in SEVR at the 15th, 20th and 25th minutes of the operation
  From the derived central aortic pulse pressure, calculations can be made, using the area under the systolic and diastolic part of the curve.

CONTACTS AND LOCATIONS:
Overall Officials: Csilla Molnár, MD, PhD, Principal Investigator — University of Debrecen Medical and Health Science Center Department of Anesthesiology and Intensive Care 4032-Debrecen, Nagyerdei krt 98. Hungary Tel/fax: +36-52-255-347
Locations (1):
- University of Debrecen Medical and Health Science Center Department of Anesthesiology and Intensive Care, Debrecen, Hungary

REFERENCES:
- [Result] Fulesdi B, Limburg M, Bereczki D, Kaplar M, Molnar C, Kappelmayer J, Neuwirth G, Csiba L. Cerebrovascular reactivity and reserve capacity in type II diabetes mellitus. J Diabetes Complications. 1999 Jul-Aug;13(4):191-9. doi: 10.1016/s1056-8727(99)00044-6. PMID 10616858
- [Result] McCulloch TJ, Thompson CL, Turner MJ. A randomized crossover comparison of the effects of propofol and sevoflurane on cerebral hemodynamics during carotid endarterectomy. Anesthesiology. 2007 Jan;106(1):56-64. doi: 10.1097/00000542-200701000-00012. PMID 17197845
- [Result] Lan YC, Shen CH, Kang HM, Chong FC. Pulse transit time reveals drug kinetics on vascular changes affected by propofol. Comput Methods Biomech Biomed Engin. 2012;15(9):949-52. doi: 10.1080/10255842.2011.567981. Epub 2011 May 24. PMID 21547779
- [Result] Strebel S, Kaufmann M, Guardiola PM, Schaefer HG. Cerebral vasomotor responsiveness to carbon dioxide is preserved during propofol and midazolam anesthesia in humans. Anesth Analg. 1994 May;78(5):884-8. doi: 10.1213/00000539-199405000-00009. PMID 8160985
- [Result] Holzer A, Winter W, Greher M, Reddy M, Stark J, Donner A, Zimpfer M, Illievich UM. A comparison of propofol and sevoflurane anaesthesia: effects on aortic blood flow velocity and middle cerebral artery blood flow velocity. Anaesthesia. 2003 Mar;58(3):217-22. doi: 10.1046/j.1365-2044.2003.03041.x. PMID 12603451
- [Result] Previgliano IJ. Assessment: transcranial Doppler ultrasonography: report of the Therapeutics and Technology Assessment Subcommittee of the American Academy of Neurology. Neurology. 2004 Dec 28;63(12):2457-8; author reply 2457-8. No abstract available. PMID 15630765
- [Derived] Juhasz M, Pall D, Fulesdi B, Molnar L, Vegh T, Molnar C. The effect of propofol-sufentanil intravenous anesthesia on systemic and cerebral circulation, cerebral autoregulation and CO2 reactivity: a case series. Braz J Anesthesiol. 2021 Sep-Oct;71(5):558-564. doi: 10.1016/j.bjane.2021.04.002. Epub 2021 Apr 23. PMID 33901551